CLINICAL TRIAL: NCT02994069
Title: Comparison of Every 3 Week Versus Weekly Cisplatin Concurrent With Radiation in Squamous Cell Carcinoma of the Head and Neck (SCCHN) and Correlation With Oxidative Stress Markers
Brief Title: Cisplatin + Radiation in SCCHN and Correlation With Oxidative Stress Markers
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Susanne Arnold (Other)
Responsible Party: Sponsor-Investigator, Susanne Arnold, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16-HN-29
Record Dates: First submitted 2016-12-12; First posted 2016-12-15 (Estimated); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Carcinoma, Squamous Cell; Head and Neck Cancer
Keywords: Cisplatin; Squamous Cell; Carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell; Head and Neck Neoplasms; Carcinoma | interventions — Cisplatin; Drug Therapy

STUDY DESIGN:
Masking Description: Unblinded trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Every 3 Weeks Cisplatin + XRT (Experimental): Every 3 Weeks Cisplatin + XRT
  Interventions: Drug: Cisplatin; Radiation: XRT
- Weekly Cisplatin + XRT (Experimental): Weekly Cisplatin + XRT
  Interventions: Drug: Cisplatin; Radiation: XRT

INTERVENTIONS:
Drug: Cisplatin — Cisplatin
  Other Names: chemotherapy
Radiation: XRT — Radiation Therapy

SUMMARY:
Patients will receive standard of care radiation therapy to the primary tumor of the head and neck and involved nodal metastasis and draining nodal basin and either weekly cisplatin or every 3-week cisplatin in locally advanced SCCHN. The relationship between cisplatin toxicity and the level of reactive oxygen species generated by the drug in subjects with squamous cell carcinoma of the head and neck treated on this trial.

DETAILED DESCRIPTION:
Patients will first be designated as either: a) Cohort 1 (locally advanced non-nasopharyngeal SCCHN that is unresectable) OR b) Cohort 2 (resected and at high risk of recurrence with at least one of the following criteria: extracapsular nodal extension, or invasive cancer at the primary tumor resection margin (positive margin), lymphovascular invasion or perineural invasion, pT3 or pT4 primary, or the presence of multilevel nodal disease. Subjects will then be randomized to receive either Arm 1 or Arm 2 cisplatin.

Radiation and Cisplatin will be given concurrently and should start on the same day, ±1 day. Radiation will continue without interruption whenever possible.

Treatment will consist of standard of care radiation therapy to the primary tumor of the head and neck and involved nodal metastasis and draining nodal basin, as determined by treating radiation oncologist. Patients will be randomized to receive cisplatin at 100 mg/m2 every 3 weeks (3 doses) during radiation versus cisplatin at 40 mg/m2 once weekly (7 doses) during radiation. This will provide similar cumulative doses of cisplatin in all arms of the study.IMRT will be delivered in 30-35 fractions over 6-7 weeks, 5 fractions weekly.

In the absence of treatment delays due to adverse event(s), treatment will continue for 7 weeks or until one of the following criteria applies:

Disease progression,Intercurrent illness that prevents further administration of treatment, Unacceptable adverse event(s), Patient decides to withdraw from the study, or General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator.

Patients will be followed for 2 years after completion of chemoradiation or until death, whichever occurs first, for toxicity and PFS.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically (histologically or cytologically) proven diagnosis of head and neck squamous cell carcinoma (HNSCC) involving the oral cavity, oropharynx, larynx, hypopharynx, paranasal sinuses or unknown primary squamous carcinoma limited to the head and neck region. Cohort 1: Unresectable locally advanced non-nasopharyngeal SCCHN without evidence of distant metastases. Cohort 2: Patients with non-nasopharyngeal SCCHN who have undergone gross total surgical resection within 63 days prior to registration. Patients must have at least 1 of the following high-risk pathologic features: extracapsular nodal extension, invasive cancer at the primary tumor resection margin (positive margin), lymphovascular invasion or perineural invasion, or the presence of multilevel nodal disease. Patients must be without evidence of distant metastases.
* Women of childbearing potential and male participants who are sexually active must agree to use a medically effective means of birth control.
* Cohort 1: Patients in Cohort 1 must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as ≥ 20 mm (≥ 2 cm) with conventional techniques or as ≥ 10 mm (≥ 1 cm) with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease. Cohort 2: Subjects in the post-operative setting (Cohort 2) are not required to have measurable disease and response rate will not be assessed in cohort 2.
* Patients may have a history of prior head and neck malignancy, but must be able to tolerate full dose radiation and chemotherapy for the current head and neck cancer, as determined by the treating oncologist.
* Age ≥18 years.
* ECOG performance status 0, 1 or 2
* Life expectancy of greater than 12 weeks.
* Patients must have normal organ and marrow function assessed within 14 days prior to registration as defined below: absolute neutrophil count ≥1,000/mcL, platelets ≥100,000/mcL, creatinine within normal institutional limits OR creatinine clearance ≥60 mL/min/1.73 m2 (for patients with creatinine levels above institutional normal).
* No prior chemotherapy for the current locally advanced SCCHN is allowed. Prior radiation or chemotherapy for a previous head and neck cancer is allowed provided full dose cisplatin and radiation can be delivered to the patient in this clinical trial and provided the patient is in remission from the prior head and neck cancer, and can undergo full dose radiation and chemotherapy for the current primary head and neck cancer.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, throughout the duration of active treatment and for 4 months after completion of chemotherapy and radiation.
* Cisplatin and radiation are known teratogens. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, throughout the duration of active treatment and for 4 months after completion of chemotherapy and radiation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of active study treatment, and for 4 months after completion of chemotherapy and radiation (both induction and definitive) administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients who are receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cisplatin.
* Patients with greater than grade 2 hearing loss.
* No other prior malignancy is allowed except for the following: head and neck cancer in remission, adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated previous Stage I or II cancer from which the patient is currently in complete remission or other cancer from which the patient has been disease-free for 2 years.
* Patients with nasopharynx or salivary gland primary site.
* Patients with distant metastatic disease (M1c) from the current head and neck cancer including brain metastasis.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (grade 3 or greater), symptomatic congestive heart failure, unstable angina pectoris, symptomatic cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Subjects with significant symptoms of congestive heart failure who would not be expected to tolerate the IV hydration for cisplatin are excluded.
* Pregnant women are excluded from this study because cisplatin and radiation are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cisplatin and radiation, breastfeeding should be discontinued if the mother is treated with cisplatin or radiation on this trial.
* HIV-positive patients with uncontrolled HIV despite combination antiretroviral therapy are ineligible because of the potential for increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2029-10-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Arnold, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Every 3 Weeks Cisplatin + XRT | Weekly Cisplatin + XRT
Started | 39 | 41
Cohort 1 | 30 | 32
Cohort 2 | 9 | 9
Completed | 24 | 22
Not Completed | 15 | 19
Not completed — Death | 7 | 13
Not completed — Adverse Event | 1 | 0
Not completed — Other | 2 | 0
Not completed — still on follow up/treatment | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Every 3 Weeks Cisplatin + XRT | Weekly Cisplatin + XRT | Total
Number analyzed (Participants) | 39 | 41 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.26 (9.33) | 59.07 (8.23) | 57.7 (8.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 27 | 30 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 38 | 40 | 78
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 35 | 38 | 73
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 39 | 41 | 80

OUTCOME MEASURES:

1. Primary Outcome: CTCAE Grade 3-5 Cisplatin-related Adverse Event Rate (Percentage)
Description: Rate of grade 3-5 cisplatin-related adverse events expressed as a percentage of each cohort of patients occurring within 90 days of initiation of concurrent radiation and chemotherapy; Rate calculated from number of patients with at least one cisplatin-related AEs with grade 3-5 within 90 days of the 1st treatment. This primary endpoint is the percentage of subjects experiencing cisplatin-related actual toxicities in each group estimated along with exact 95% binomial confidence intervals.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Every 3 Weeks Cisplatin + XRT | Weekly Cisplatin + XRT
Number analyzed (Participants) | 39 | 41
percentage of participants | 74.36 (6.99) | 68.29 (7.27)

2. Secondary Outcome: Local Control Rates
Description: 2 year local control rate
Time Frame: 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Survival
Description: Overall survival
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Every 3 Weeks Cisplatin + XRT | Weekly Cisplatin + XRT
Number analyzed (Participants) | 39 | 41
days | 687.5 (10.45) | 517.06 (14.71)

ADVERSE EVENTS:
Time Frame: 2 years
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting; Grade 3 or higher treatment related Adverse Events are listed as serious adverse events
Arm/Group | Every 3 Weeks Cisplatin + XRT | Weekly Cisplatin + XRT
All-Cause Mortality (participants affected / at risk) | 7/39 | 13/41
Serious Adverse Events (participants affected / at risk) | 39/39 | 41/41
Other Adverse Events (participants affected / at risk) | 8/39 | 10/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Every 3 Weeks Cisplatin + XRT (N=39) | Weekly Cisplatin + XRT (N=41)
Anemia (Blood and lymphatic system disorders) | 1 | 3
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 4
Other (Blood and lymphatic system disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 5 | 1
Dysphagia (Gastrointestinal disorders) | 7 | 4
Mucositis Oral (Gastrointestinal disorders) | 11 | 15
Nausea (Gastrointestinal disorders) | 10 | 2
Vomiting (Gastrointestinal disorders) | 11 | 3
Oral Pain (Gastrointestinal disorders) | 1 | 13
Fatigue (General disorders) | 1 | 3
Sinusitis (Infections and infestations) | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 1
Esophagitis (Gastrointestinal disorders) | 0 | 1
pain (General disorders) | 0 | 1
Bronchial Infection (Infections and infestations) | 0 | 1
Mucosal Infection (Infections and infestations) | 0 | 1
Other (Infections and infestations) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 1
Weight loss (Investigations) | 0 | 1
White blood cell decreased (Investigations) | 10 | 12
Lymphocyte count decreased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 8 | 2
CD4 lymphocytes decreased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 3
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Other (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 1
Hematuria (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Every 3 Weeks Cisplatin + XRT (N=39) | Weekly Cisplatin + XRT (N=41)
Other (Blood and lymphatic system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 2 | 1
Oral dysesthesia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT02994069/Prot_SAP_000.pdf